CLINICAL TRIAL: NCT00319124
Title: Evaluation of Function and Effect of Exercise in Patients With Osteoarthritis of the Hip.A Case-control Study.
Brief Title: Exercise Therapy and Patient Education for Individuals With Hip Osteoarthritis of the Hip. A Case-Control Study
Status: Completed | Type: Observational
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Norwegian Foundation for Health and Rehabilitation (Other)
Responsible Party: Principal Investigator, May Arna Risberg, Professor, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Other Study IDs: 03b-2005-NAR
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2016-03-02 (Estimated); Status verified 2012-05

CONDITIONS: Hip Osteoarthritis
Keywords: Hip Osteoarthritis, muscle strength, range of motion, aerobic capacity, functional capacity, health-related quality of life
MeSH Terms: conditions — Osteoarthritis, Hip

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case: Patients with hip Osteoarthritis
- Control: Healthy controls without hip osteoarthritis

SUMMARY:
To identify differences between patients with OA of the hip in an early stage and a healthy control group.

Hypothesis 1.1 There are significant differences between patients with OA of the hip in an early stage and a healthy control group in terms of functional capacity, biomechanical / kinematic variables, muscle strength and range of motion.

Osteoarthritis (OA) is by far the most prevalent joint disorder today. The knee and the hip are large joints to be targeted and is an important cause of pain and disability. In knee OA, it is shown that significant risk factors in developing the disease are quadriceps weakness, joint instability, and changes in joint loading. A few studies on hip OA have shown altered gait pattern, which affect joint loading, and one study has shown weakness in abductors, adductors and flexors around the hip. As joint loading and muscle weakness are important factors in the development in knee OA, it might as well be factors influencing OA in the hip. The purpose of this case-control studies was to compare hip OA patients to a healthy control group regarding biomechanical and clinical differences. Patients with hip pain, activity limitations (Harris Hip Score 60-95 p) and radiographically verified hip OA was included. The healthy control group will have a Harris Hip Score of 100 p. One hundred and ten patients and fifty controls will be asked to fill in questionnaires on pain, stiffness and physical function (WOMAC), quality-of-life (SF-36 v2), self-efficacy (Lorigue), and activity (PASE) in addition to perform 6-minute walk test, sub-maximal cardiovascular function, strength, and hip range of motion tests. Additionally, Qualisys Pro reflex 3D motion analysis system will be used during walking, one-leg standing, and raising from a chair on a sub-group of 40 patients and 20 controls.

DETAILED DESCRIPTION:
Aim 1 To identify differences between patients with OA of the hip in an early stage and a healthy control group.

Hypothesis 1.1 There are significant differences between patients with OA of the hip in an early stage and a healthy control group in terms of functional capacity, biomechanical / kinematic variables, muscle strength and range of motion.

Material and methods.

Design. A case-control study

Inclusion / exclusion criteria. Twenty-five patients diagnosed with unilateral or bilateral OA of the hip will be recruited from the Norwegian Sport Medicine Centre, Diakonhjemmet and from the Orthopaedic Centre, Ullevål University Hospital, Oslo, Norway. PPatients will also be recruited through ads in newspaper and brief information in national tv. Radiographiccally verified OA of the hip will be in accordance with Danielsson's criteria for minimal joint space. Patients will be excluded if they have a history of resent trauma or functional impairment to the lower limbs or diseases which might interfere with participation.

Control subjects will have no health problems and no injuries or functional impairment to the lower limbs and will be matched to the patients with OA of the hip by age and gender.

Outcome measures.

Background descriptive data, including anthropometrical (age, gender, height, weight) and sociodemographic information (marital status, social support, leisure time, sick-leave, physical activity, occupational background, co-morbidity, hip pain history, former treatment for hip pain / OA), and consumption of analgetics will be collected by questionnaire at inclusion. Outcome measures will cover all functional levels defined by the World Health Organization's (WHO) International Classification of Functioning, Disability, and Health (2002) and will include:

Pain and activity limitation: Hip pain will be assessed by a horizontal visual analogue scale (VAS) (0-100 mm; 0 represents "no pain" and 100 represents "as much pain he/she can possibly imagine") (Revill et al. 1976). Both self-reported and observed functional capacity will be evaluated. Self-reported functional capacity will be registered by the disease-specific questionnaire Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) (Bellamy et al. 1988). Observed functional capacity will be assessed by the 6 minute walking test (Enright, 2003), where the patient is instructed to walk as quickly/fast as possible forth and back on a 20 m course, and by the subaximal bikecycle test (Astrand, 1986) where the heart-rate is registered on a constant load and speed.

Health related quality of life and pain management: Quality of life will be assessed by using the generic questionnaire SF-36 v.2 (Jenkinson, 1999). Self-efficacy beliefs for pain will be registered using the self-efficacy subscale for controlling pain developed by Lorig et al (Lorig et al. 1989). The scale is found to be valid and reproducible in patients with chronic arthritis (Lorig et al. 1989).

Gait analysis: Kinematic data will be collected using Qualisys pro-reflex motion analysis system with eight cameras at a sampling frequency of 240 Hz and synchronized with two force platforms sampling at a rate of 960Hz (AMTI Model LG6). All markers will be present during standing calibration. During the dynamic trials all the anatomical markers will be removed.

Subjects will be instructed to walk along a 17m walkway in which two force plates are embedded. The subjects will walk at their self-selected pace and practice trials will be performed until the subject could contact the force platforms with only one foot (not targeting) and with a constant velocity within 5% deviation. Speed will be measured by photoelectric beams located 3.06m apart, midway along the walkway. Experienced physical therapists will be responsible for patient information, instruction and data collection.

Muscle strength: Muscle strength of hip extensors, -flexors, knee flexors and -extensors, and ankle flexors and extensors, in addition to ankle plantar flexion will be tested isokinetically according to the manufacturer's manual (Cybex 6000). Isokinetic muscle testing is commonly used in the literature in various patient populations (Inkster et al. 2003; Holm et al. 2000b; Brox et al. 1995; Lephart et al. 1993; Newton et al. 1993). The test protocol will consist of five repetitions at an angular velocity of 60 deg/sec at maximal performance. In order to prepare patients for the test, eliminate learning effects and to obtain stable performance, patients will be given four test-repetitions at the same speed before the main test. An experienced physical therapist will perform the test.

Range of motion: Range of motion will be measured by goniometer according to standard procedures (Holm et al. 2000a).

Follow up: Data will be collected at inclusion (patients and control subjects) and after the intervention period (patients).

Blinding: Personnel responsible for the intervention will not be involved in data collection.

Registration of complications, drop-outs and adherence: Complications and drop-outs will be registered by persons responsible for data collection. Adherence to the exercise protocol will be registered by the physical therapists responsible for the treatment.

Power calculations: Lack of information from studies of comparable OA populations in the literature makes it difficult to make precise power calculations. Assumption of sample size (110 patients and 50 control subjects) is therefore based on results from former studies in patients with OA of the knee or mixed populations of knee- and hip patients.

Statistical analysis: Both non-parametric and parametric statistics will be used for data analysis.

Ethics: All patients and control subjects will receive written and oral information about the study and sign an informed consent before inclusion (enclosed). The project will be performed according to recommendations of the Helsinki Declaration and application will be sent to the Regional Committee of Medical Research Ethics in Oslo in November 2003.

ELIGIBILITY:
Inclusion Criteria for patients with hip OA:

* 110 patients between 40 and 80 years old with uni- or bilateral hip disability
* Harris Hip Score (36) between 60 and 95.Harris Hip score(0-100 points) is widely used as an assessment of hip function in patients with hip OA. Harris Hip Score of 60 or below are used regularly at our institution as one of the criteria for hip surgery (arthroplasty).
* Patients will be included if they have more than 3 months of hip pain.
* Patients with radiographic verified hip OA (Danielson's criteria for radiographic OA: Danielsson's criteria for minimal joint space: <4 mm <70 years, <3 mm ≥70 years, or 1 mm difference between hips).
* Fifty control subjects will have no health problems and no injuries or functional impairment to the lower limbs and will be matched to the patients with OA of the hip by age and gender.

Exclusion Criteria:

* Patients have a history of resent trauma or functional impairment to the lower limbs or diseases which might interfere with participation (rheumatoid arthritis, cancer, osteoporosis, severe back pain, knee OA).
* Patients with co-morbidities not tolerating physical activities

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with hip osteoarthritis and mild to moderate pain. Matched controls with no hip pain.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2005-04; Primary Completion 2008-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index(WOMAC) | Baseline

SECONDARY OUTCOMES:
SF-36 (quality of life) | Baseline
PASE (activity score) | Baseline
muscle strength tests (Cybex 6000) | Baseline
gait analysis (biomechanical analysis) | Baseline
6 minutes walking test | Baseline
Åstrand's bike test | Baseline
Range of Motion (goniometer) | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: May Arna Risberg, PT,PhD, Principal Investigator — NAR-Department of Orthopaedics, Oslo University Hospital
Locations (1):
- NAR- Department of Orthopaedics, Oslo University Hospital & Hjelp24NIMI, Oslo, Oslo County, Norway

REFERENCES:
- [Result] Rydevik K, Fernandes L, Nordsletten L, Risberg MA. Functioning and disability in patients with hip osteoarthritis with mild to moderate pain. J Orthop Sports Phys Ther. 2010 Oct;40(10):616-24. doi: 10.2519/jospt.2010.3346. PMID 20811166
- [Result] Eitzen I, Fernandes L, Nordsletten L, Risberg MA. Sagittal plane gait characteristics in hip osteoarthritis patients with mild to moderate symptoms compared to healthy controls: a cross-sectional study. BMC Musculoskelet Disord. 2012 Dec 20;13:258. doi: 10.1186/1471-2474-13-258. PMID 23256709
- See also: Related Info — http://www.active-rehab.no